CLINICAL TRIAL: NCT07358962
Title: Mild Cognitive Impairment and Psychopathology: Effects on Awareness, Social Life, and Work. Cross-sectional Observational Study
Brief Title: Mild Cognitive Impairment and Psychopathology
Acronym: MIND
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Irene Cappadona, PSYCHOLOGIST, IRCCS Centro Neurolesi Bonino Pulejo
Other Study IDs: 11/2025
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Mild Cognitive Impairment (MCI); Psychopathological disorders; Anosognosia; Cognitive decline; Social functioning; Work functioning; Neuropsychological assessment
MeSH Terms: conditions — Cognitive Dysfunction; Agnosia; Social Adjustment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MCI: Patients diagnosed with Mild Cognitive Impairment

SUMMARY:
Mild Cognitive Impairment (MCI) is a condition characterized by cognitive deterioration greater than what is expected from normal aging, representing an important risk factor for the development of dementia. Early assessment of cognitive functions is therefore essential for promptly identifying any signs of decline. In addition to cognitive aspects, it is equally important to consider the possible psychopathological profile of patients, as such disorders can significantly influence the progression of the disease, quality of life, and the ability to manage daily activities. This protocol aims to explore the presence of psychopathological disorders in patients with MCI, with particular attention to their impact on awareness of cognitive deficits (anosognosia) and on the subjective perception of difficulties in daily life, especially in social and work contexts. The study seeks to outline a comprehensive picture of the psychopathological profile in patients with MCI, facilitating the identification of targeted and personalized interventions capable of improving clinical management and the overall well-being of the individual.

DETAILED DESCRIPTION:
The study has a cross-sectional observational design, with data collected at a single time point (T0). The overall duration of the study, estimated at approximately 12 months, will depend on the time required to complete participant enrollment, data analysis, and dissemination of results. The purpose of this protocol is to investigate the presence of psychopathological disorders in patients with Mild Cognitive Impairment (MCI), with particular attention to their impact on awareness of cognitive deficits (anosognosia) and on the ability to cope with difficulties in social and work-related activities.

In this context, the study aims to outline a broader and more structured picture of the psychopathological profile of patients with MCI. This perspective will make it possible to analyze the interactions between emotional aspects, personality characteristics, and cognitive decline, with the goal of identifying more targeted and personalized intervention strategies capable of improving clinical management and promoting overall well-being.

The primary objective is to assess the presence of psychopathological disorders in patients with Mild Cognitive Impairment (MCI). The secondary objectives are to examine the impact of psychopathological disorders on the level of awareness of one's cognitive decline (partial or total anosognosia) and to evaluate how such disorders affect daily life by comparing the subjective perception of difficulties in social and work contexts.

As this is a cross-sectional observational study involving a single group of MCI patients, the sample size was estimated a priori using G*Power 3.1 with a one-sample binomial test (two-tailed) for the primary objective, the estimation of the prevalence of psychopathological disorders. Based on the literature, an expected prevalence of p1 = 0.20 was assumed, to be compared with a reference value of p2 = 0.32 (α = 0.05; power 1-β = 0.85), resulting in an estimated sample size of N = 118 subjects. Considering a 15% margin for possible drop-outs or invalid data, the final sample size was set at N = 136 participants.

Subjects will be included in the study if, based on available clinical documentation, they meet the following requirements: age between 50 and 72 years; diagnosis of Mild Cognitive Impairment (MCI), referred to the Neuropsychology Clinic for an initial evaluation or clinical follow-up; absence of behavioral, psychiatric, or sensory disorders severe enough to significantly compromise the performance of cognitive tests or the completion of questionnaires.

Subjects will be excluded from the study if clinical documentation reveals at least one of the following conditions: neurological disorders other than MCI, such as recent stroke, severe traumatic brain injury, epilepsy, multiple sclerosis, or other atypical neurodegenerative diseases; major psychiatric comorbidities not stabilized at the time of assessment (e.g., schizophrenia, bipolar disorder in an active phase, untreated severe depression); severe uncorrected sensory deficits (visual or auditory) that could compromise the validity of cognitive and functional assessments; use of medications with significant potential cognitive impact (e.g., sedatives, high-dose antipsychotics) not stabilized at the time of evaluation; terminal-stage internal or oncological diseases, or other medical conditions that significantly interfere with the performance of assessment procedures.

Each patient deemed eligible for the study will be informed about the study's purpose and will freely decide whether to participate. Only after the patient, or their Legal Representative, has agreed to participate in the study and signed the informed consent form may the Investigator proceed with the planned procedures.

The patient's pathway through the study will proceed as follows: clinical data for each subject will be shared through a secure database accessible to study collaborators using personal credentials. After verifying inclusion and exclusion criteria and obtaining informed consent, patients will proceed to the subsequent phases of the study.

1. Enrollment phase: verification of inclusion and exclusion criteria; collection of demographic data; collection of the subject's clinical history.
2. Assessment phase: eligible patients will undergo a battery of standardized tests aimed at assessing cognitive functioning, the presence of psychopathological traits, subjective awareness of deficits, and personal perception and ability to manage difficulties in daily activities. The battery will include the following instruments: Brief Cognitive Status Examination (BCSE) and/or Montreal Cognitive Assessment (MoCA), Minnesota Multiphasic Personality Inventory-3 (MMPI-3), Beck Depression Inventory (BDI-II), State-Trait Anxiety Inventory (STAI-Y), Cognitive Failures Questionnaire (CFQ), Social Functioning Questionnaire (SFQ), Instrumental Activities of Daily Living (IADL).

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 72 years;
* Diagnosis of Mild Cognitive Impairment (MCI), with referral to the Neuropsychology clinic for an initial evaluation or for clinical monitoring;
* Absence of behavioral, psychiatric, or sensory disorders that could significantly compromise the performance of cognitive tests or the completion of questionnaires.

Exclusion Criteria:

* Neurological disorders other than MCI, such as recent stroke, severe traumatic brain injury, epilepsy, multiple sclerosis, or other atypical neurodegenerative diseases;
* Major psychiatric comorbidities not stabilized at the time of the assessment (e.g., schizophrenia, bipolar disorder in an active phase, untreated severe depression);
* Severe uncorrected sensory deficits (visual or hearing) capable of compromising the validity of cognitive and functional assessments;
* Use of medications with significant potential cognitive impact (e.g., sedatives, high-dose antipsychotics) not stabilized at the time of the assessment;
* Terminal-stage internal or oncological diseases, or other medical conditions that significantly interfere with the assessment procedures.

Ages: 50 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As this is a cross-sectional observational study involving a single group of MCI patients, the sample size was estimated a priori using G*Power 3.1 with a one-sample binomial test (two-tailed) for the primary objective, namely the estimation of the prevalence of psychopathological disorders. In accordance with the literature, an expected prevalence of p1 = 0.20 was assumed and compared with a reference value of p2 = 0.32 (α = 0.05; power 1-β = 0.85), yielding an estimated sample size of N = 118 subjects. Considering a 15% margin for potential drop-outs or invalid data, the final sample size was set at N = 136 participants.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-01-12 (Estimated); Study Completion 2027-01-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of psychopathological disorders in patients with MCI | 12 months
  The primary outcome variable is the presence of psychopathological disorders, assessed using the MMPI-3 test, which is used as an indicator of the psychopathological profile in patients with mild cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Centro Neurolesi Bonino Pulejo, Messina, Me, Italy

IPD SHARING:
Plan to Share IPD: No